CLINICAL TRIAL: NCT01642693
Title: Histological Changes of The Dentinal-Pulp Complex and Root Resorption in Maxillary Premolars With Intrusive Orthodontic Movements Under a Low Power Laser Effect
Brief Title: Histological Change of The Dentinal-Pulp Complex and Root Resorption
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Paula Villa M, Partial time proffesor in Endodontics, Universidad de Antioquia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2006-007
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Laser; Intrusion; Histology; Resorption
Keywords: root resorption; low-power laser; orthodontic tooth movement; pulp changes
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Teeth with intrusive movement and low power laser (Experimental): Histological changes and root resorption were assesed in Teeth with intrusive movement after a low power laser application
  Interventions: Radiation: Low power laser in teeth after intrusive movement
- Teeth with intrusive movements with no laser (Experimental): Histological changes and root resorption in Teeth with intrusive movements with no laser
  Interventions: Other: Simulated laser in teeth with intrusive movements

INTERVENTIONS:
Radiation: Low power laser in teeth after intrusive movement — Low power laser was aplied to premolar teeth under an intrusive movement to study histological changes and root resorption
  Arms: Teeth with intrusive movement and low power laser
Other: Simulated laser in teeth with intrusive movements — Simulated laser in teeth with intrusive movements for histological and root resorption changes
  Arms: Teeth with intrusive movements with no laser

SUMMARY:
The purpose of the study is evaluate the histological changes of the dentinal-pulp complex and root resorption in maxillary premolars with intrusive orthodontic movement under a low power laser effects.

DETAILED DESCRIPTION:
Orthodontics movements can cause inflamatory changes in the pulp and external inflamatory root resorption, different methods have been suggested to control that changes as the use of the low power laser. The objective of this study is to evaluate the low power laser effect on the inflamatory pulpar change and inflamatory external root resorption in maxillary premolars with intrusive orthodontic movements of 4 ounces during 12 weeks. Total sample were 34 healthy teeth, 16 were used to evaluate the normal standar and 18 were divided in two groups, the experimental group with the low power laser effect had a dose of 18 joules after activations of the orthodontic intrusion and the control group had a simulated effect in the same orthodontic movement. Teeth were extacted after 12 weeks and histological changes were evaluated in the dentinal-pulp complex and the pesence of external inflamatory root resorption. Findins suggest that low power. Laser decreased the inflamatory changes of the dentinal - pulp complex and the severity of the external inflamatory root resorption.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first premolar extraction indicated
* Patients with no sistemic diseases
* Healthy premolars with completed root and no trauma or restoration

Exclusion Criteria:

* Sistemics diseased
* Restoration, trauma in first premolars
* root uncompleted

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Teeth with intrusive movement and low power laser | 12 weeks
  Histological changes and root resorption were assesed in Teeth with intrusive movement after a low power laser application

SECONDARY OUTCOMES:
Teeth with intrusive movements with no laser exposition | 12 weeks
  Histological changes and root resorption were assesed in Teeth with intrusive movement with no laser exposition

CONTACTS AND LOCATIONS:
Locations (1):
- Paula Villa M, Medellín, Antioquia, Colombia

REFERENCES:
- See also: Related Info — http://www.udea.edu.co